CLINICAL TRIAL: NCT03881592
Title: A Czech Pharmaco-epidemiological Real-World Data Study Focused on CLL Patient Treatment Options and Their Effectiveness
Brief Title: Real-World Data Study Focused on Chronic Lymphocytic Leukemia (CLL) Patient Treatment Options and Their Effectiveness
Acronym: GO-CLLEAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Michael Doubek, M.D., Ph.D, Head of the Czech CLL Study Group, Brno University Hospital
Other Study IDs: ML41010
Record Dates: First submitted 2019-03-03; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- R-Clb patients: Patients treated with the combination of Rituximab + chlorambucil
- R-B patients: Patients treated with the combination of Rituximab + bendamustine
- Obi-Clb patients: Patients treated with the combination of Obinutuzumab + chlorambucil

SUMMARY:
This study will be a secondary use of data, focusing on patients treated with combination therapy Obi-Clb, R-Clb or R-B, in a non-interventional, open label, national, multicenter setting. Retrospective analysis of data coming from registry database CLLEAR (www.leukemia-cell.org )that capture data on clinical and treatment practices in CLL. Data will be retrospectively analyzed.

DETAILED DESCRIPTION:
This study will be a secondary use of data, focusing on patients treated with various treatment regimens (including obinutuzumab based regimen) used in the Czech Republic in a non-interventional, open label, national, multicenter setting. Retrospective analysis of data coming from registry database CLLEAR that capture data on clinical and treatment practices in CLL. This study is not a face to face analysis of treatment regimens. The results of this study could be used to compare with the results from other studies.

Analytical population, selection criteria and sample size

All CLL patients diagnosed, treated or followed in seven leading hematology centers in the Czech Republic since 2011 onward are included in the CLLEAR registry; there are no exclusion criteria. These centers include University Hospital (UH) Brno, General Faculty Hospital in Prague, University Hospital Hradec Kralove, University Hospital Olomouc, University Hospital Ostrava, University Hospital Plzen and Oncology Center Novy Jicin.

In this study, all patients treated with Obi-Clb, R-B and R-Clb regimens and included into the CLLEAR database will be analyzed. There no other selection criteria.

It is estimated that 400 patients will be analyzed in the study.

Primary and secondary objectives

General To assess effectiveness and disability accrual in Czech CLL patients treated with various treatment regimens in similar demographic population using available real-world data from the CLLEAR registry. The results of this study could be used to compare with the results from other studies.

Primary objective

1. Patients 'profile - Patients´ demographic characteristics such as age, gender, occurrence of comorbidities, level of Cumulative Illness Rating Scale (CIRS score), renal function etc. in patients treated with various treatment regimens (Obinutuzumab+chlorambucil (Obi-Clb), rituximab+chlorambucil (R-Clb), rituximab+bendamustin (R-B)).
2. Effectiveness of the treatment regimens (Obi-Clb, R-Clb, R-B) in patients with above defined demographic characteristics based on measured parameters as indication/direct correlation of effectiveness - overall response rate (ORR), complete response (CR), Progression-free Survival (PFS), Minimal Residual Disease (MRD) negativity.

Secondary objectives

The secondary objectives of this study are as follows:

1. The frequency (in %) of both hematologic adverse events (neutropenia, thrombocytopenia) and non-hematologic (grade ≥3 infections and Infusion Related Reaction - IRRs) in patient population.
2. The frequency of comorbidities in patient population.
3. The need for treatment adjustment (e.g. decreases in number of cycles) in patients.
4. The percentage of adverse events (infections) in above defined patient population requiring hospitalization.

Data protection and data monitoring

All data will be analyzed from the CLLEAR registry. Personal data protection and implementation of appropriate legislation regarding personal data protection (GDPR) is dealt with within registry CLLEAR. In the database CLLEAR, there are strict rules on the protection of personal data due to Czech law.

All patients' data are anonymized. All patients have to sign informed consent. The registry was approved by multicentric ethics committee. It is an incremental data set that is updated periodically, every 6 months, and regularly validated by an independent central data manager. No monitoring of centers is performed.

Regulatory and legislative requirements

General Informed Consent is not part of this study as this study uses data from separate registry CLLEAR. Registry has its own Informed Consents. Informed consent based essentially on the data privacy clause is obtained from each patient prior to data collection into the registry CLLEAR as two original documents signed by the patient. One original Informed Consent Form (ICF) is filed with the patient´s documentation in the clinical center and the second original ICF is given to the patient.

This is a non-interventional post-registration study that must follow all local law or regulations and medical practice. Local legislative requirements of the Czech Republic will be applied.

Quality assurance and control

The project will be carried in accordance with IBA (Institute of Biostatistics and Analyses) internal quality management system and procedures (established Quality Management System according to the norm of the International Organization for Standardization - ISO 9001:2012 including the quality manual; system Information technology according to ISO/IEC 20000-1:2012).

Study data analysis

This study is secondary data use, observational, with data and analysis gathered as indicated in the following sections.

The following general /baseline and therapeutic characteristics and measures will be collected: age, gender, comorbidities, level of CIRS score, renal function (e.g. creatinine level), side effects hematology related and unrelated and the need for hospitalization, number of chemotherapeutic cycles, response to treatment (i.e. complete or partial remission), occurrence of progression and presence of minimal residual disease (MRD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Lymphocytic Leukemia
* Patients treated with Bendamustin plus Rituximab, Rituximab plus Chlorambucil or Obinutuzumab plus Chlorambucil regimens as first line of treatment
* Provision of informed consent for recording of patient data in the CLLEAR registry

Exclusion Criteria:

* All untreated patients
* Patients with both Rituximab plus Chlorambucil and Bendamustin plus Rituximab or Obinutuzumab plus Chlorambucil in second or subsequent lines
* Patients with prednisone alongside analysed regimens in the first line of treatment
* Patients with RCD (Rituximab, Cyclophosphamide, Dexamethasone) or FCR (Fludarabine, Cyclophosphamide, Rituximab) or other regimen before analysed regimens within the first line of treatment
* Patients with R-Dex (Rituximab and Dexamethasone) cycles in between R-Clb cycles

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from the registry.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the treatment administration until the disease progression, death or date of data export (up to 96 months)
  PFS is defined as the number of months from the start of treatment with analyzed therapies (Obi-Clb, R-Clb, BR) until the first documentation of disease progression or death due to any cause, whichever occurred first. Kaplan-Meier method was used for evaluation.
Complete response (CR) rate | From the treatment administration up to approximately 2 months after the end of the analyzed treatment
  Complete response (remission) was assessed by using the National Cancer Institute - Working Group guidelines on CLL. It is the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. For CR definition see Hallek et al. Blood 2008 111:5446-5456; doi: https://doi.org/10.1182/blood-2007-06-093906
Partial response (PR) rate | From the treatment administration up to approximately 2 months after the end of the analyzed treatment
  Partial response (remission) was assessed by using the National Cancer Institute - Working Group guidelines on CLL. For PR definition see Hallek et al. Blood 2008 111:5446-5456; doi: https://doi.org/10.1182/blood-2007-06-093906
Overall response (ORR) rate | From the treatment administration up to approximately 2 months after the end of the analyzed treatment
  ORR is defined as the proportion of participants with complete remission (CR) or partial remission (PR) out of the total number of participants. Responses were assessed by using National Cancer Institute - Working Group guidelines on CLL.
Minimal residual disease (MRD) negativity rate | From the treatment administration up to 12 months after the end of the analyzed treatment
  The patients who achieved a CR and did not have detectable MRD in the bone marrow by four-color flow cytometry (<0.1% of cells).

SECONDARY OUTCOMES:
Frequency of patients with hematologic adverse events, non-hematologic adverse events and infusion-related reactions | From the treatment administration until the end of the analyzed treatment (up to 96 months)
  Adverse events (hematologic, non-hematologic and infusion-related reactions) were collected from the start of study treatment until the end of the treatment or end of the study. Besides the frequency of patients with a hematologic adverse event, the occurrence of neutropenia, thrombocytopenia and anaemia of different grades is presented. Beside the frequency of patients with a non-hematologic adverse event, the frequency of patients with an infection is presented.
Frequency of patients with a hematologic or non-hematologic adverse event or an infusion-related reaction that needed hospitalization | From the treatment administration until the end of the analyzed treatment (up to 96 months)
  Adverse events (hematologic, non-hematologic and infusion-related reactions) were collected from the start of study treatment until the end of the treatment or end of the study. Out of patients with at least one adverse event, the frequency of patients requiring hospitalization ir observed.
Frequency of comorbidities occurring before or during the treatment | From the date of birth of patients until the end of the analyzed treatment (up to 96 months)
  Comorbidities are defined as additional conditions co-occurring with chronic lymphocytic leukaemia. They were collected before and during the analyzed treatment.
Frequency of patients with a decrease in the number of cycles and with an increase in the number of cycles | Treatment administration (6 cycles, it means 6 months)
  A decrease in the number of cycles is when the administered number of cycles is lower than 6 (i.e. standard number of cycles) and it is considered as a treatment adjustment. An increase in the number of cycles is when the administered number of cycles is higher than 6 (i.e. standard number of cycles) and it is considered as a treatment adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Doubek, Prof,MD,PhD, Principal Investigator — The Czech CLL Study Group
Locations (2):
- Czechia (2):
  - University Hospital Brno, Department of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Hradec Králové, Department of clinical hematology, Hradec Králové

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Czech leukemia study group for life - website with the link to the CLLEAR registry — http://www.leukemia-cell.org/index-en.php?pg=cllear